CLINICAL TRIAL: NCT00805025
Title: An Open-Label, Multicenter Trial to Validate the Quality of Life Questionnaire-Bronchiectasis and to Evaluate Perception of Symptom Improvement Following One Course of Aztreonam for Inhalation Solution (AZLI) in Subjects With Bronchiectasis and Gram-negative Bacteria in the Airways
Brief Title: Evaluation of the Quality of Life Questionnaire-Bronchiectasis (QOL-B) in Patients With Bronchiectasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-219-0102
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Aztreonam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZLI (Experimental): Participants were evaluated beginning 14 days prior to starting a 28-day course of AZLI (Day 0 to Day 28), followed by post-treatment assessments every 14 days through Day 56, for a total of 70 days of participation in the study.
  Interventions: Drug: AZLI

INTERVENTIONS:
Drug: AZLI — 75 mg aztreonam for inhalation solution (AZLI), administered 3 times daily using the PARI Investigational eFlow® Nebulizer System (with a minimum of 4 hours between doses) following administration of a short-acting bronchodilator
  Other Names: Cayston®

SUMMARY:
Over the 70-day study period, eligible patients visited the study clinic every 2 weeks (total of 6 visits) and received a 28-day course of aztreonam for inhalation solution (AZLI). The Quality of Life-Bronchiectasis (QOL-B) questionnaire was completed at several time points during the study, in additional to pulmonary function testing and other standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study-related procedures
* Ability to read and understand the English language
* Bronchiectasis confirmed by CT scan of the chest
* Previous treatment with antibiotics for bronchiectasis
* Documented history of positive sputum culture for a gram-negative organism within 5 years
* Positive sputum culture for a gram-negative organism at first visit (Day -14)

Exclusion Criteria:

* Hospitalization or hemoptysis > 30 mL within 14 days of first visit (Day -14)
* Antibiotic use for respiratory symptoms within 14 days of first visit (Day -14), excluding chronic, stable azithromycin use
* Change in corticosteroid or bronchodilator regimen within 14 days of first visit (Day -14)
* Forced expiratory volume in 1 second (FEV1) < 25% predicted approximately 15 minutes following use of a bronchodilator at first visit (Day -14)
* Cigarette smoking within 6 months of first visit (Day -14)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Lamola, MD, Study Director — Gilead Sciences
Locations (24):
- United States (24):
  - Birmingham, Alabama
  - Peoria, Arizona
  - Phoenix, Arizona
  - Orange, California
  - Denver, Colorado
  - Farmington, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Olathe, Kansas
  - Boston, Massachusetts
  - Chesterfield, Missouri
  - Mineola, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Tyler, Texas
  - Charlottesville, Virginia
  - Madison, Wisconsin

REFERENCES:
- [Derived] Quittner AL, Marciel KK, Salathe MA, O'Donnell AE, Gotfried MH, Ilowite JS, Metersky ML, Flume PA, Lewis SA, McKevitt M, Montgomery AB, O'Riordan TG, Barker AF. A preliminary quality of life questionnaire-bronchiectasis: a patient-reported outcome measure for bronchiectasis. Chest. 2014 Aug;146(2):437-448. doi: 10.1378/chest.13-1891. PMID 24626872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 21 study sites in the United States. The first participant was screened on 08 December 2008. The last participant observation was on 14 October 2009.
Pre-assignment Details: 131 participants were screened and 89 were enrolled and treated.
Groups:
- AZLI: Participants were evaluated beginning 14 days prior to starting a 28-day course of aztreonam for inhalation solution (AZLI) 75 mg three times daily via investigational nebulizer (Day 0 to Day 28), followed by post-treatment assessments every 14 days through Day 56, for a total of 70 days of participation in the study.
Period: Overall Study
Arm/Group | AZLI
Started | 131
Enrolled and Treated | 89
Completed | 82
Not Completed | 49
Not completed — Screened but not enrolled/treated | 42
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Enrolled and treated participants
Groups:
- AZLI: Participants were evaluated beginning 14 days prior to starting a 28-day course of AZLI 75 mg three times daily via investigational nebulizer (Day 0 to Day 28), followed by post-treatment assessments every 14 days through Day 56, for a total of 70 days of participation in the study.
Arm/Group | AZLI
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2
  African-American | 3
  White | 84

OUTCOME MEASURES:

1. Primary Outcome: Reliability of the Respiratory Domain of the Quality of Life Questionnaire-Bronchiectasis (QOL-B)
Description: Test-retest reliability is a measure of the stability or reproducibility of a measure over a period of time during which status on the underlying construct has not changed, and is measured by the intraclass correlation of scores obtained at 2 time points within that period. Test-retest reliability of respiratory symptoms was calculated for response at Day -14 and Day 0. Reliability of the participants' QOL-B responses was assessed from an Intraclass Correlation Coefficient (ICC). A score of ≥ 0.70 would indicate strong reliability.
  The QOL-B respiratory symptoms score was transformed onto a scale of 0-100, with higher scores representing a better quality of life.
Time Frame: Day -14 to Day 0
Population: Participants who were treated and had any QOL-B measurements at both Screening and Day 0 (Visits 1 and 2) were analyzed.
Measure: Number; unit: Intraclass Correlation Coefficient
Arm/Group | AZLI
Number analyzed (Participants) | 86
Intraclass Correlation Coefficient | 0.80

2. Primary Outcome: Convergent Validity of the Respiratory Domain of the QOL-B
Description: Convergent validity was assessed at Day -14 by examining the correlations between relevant QOL-B domains and other indicators of health status: a bronchiectasis severity score based on high-resolution computerised tomography (HRCT) scan results, forced expiratory volume in 1 second (FEV1) percent predicted, 6-minute walk test (6MWT) results, and St. George's Respiratory Questionnaire (SGRQ) symptoms scores. Correlations with absolute values of 0.30 to 0.50 indicated moderate evidence of convergent validity.
Time Frame: Day -14
Population: Participants were analyzed for respiratory domain score at Day 0 against each of the other variables; those with data for both the respiratory domain score and each variable are reported.
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | AZLI
Number analyzed (Participants) | 131
Pearson correlation coefficient
  HRCT overall sentisitivity (n = 118) | -0.19
  FEV1 % predicted (n = 119) | 0.11
  6MWT (n = 121) | 0.16
  SGRQ symptoms (n = 121) | -0.75

3. Secondary Outcome: Responsiveness of the Respiratory Domain of the QOL-B as Assessed by the Anchor-based Minimal Clinically Important Difference (MCID) Following Categorization of Level of Change Using the Global Rating of Change Questionnaire (GRCQ)
Description: The anchor-based method measured the participant's perception of change at Day 28 using the GRCQ, which assesses improving/worsening symptoms. Distribution of ratings was categorized as no change (-1 to 1), minimal change (≥ 1.1 to < 3.1 or ≤ -1.1 to > -3.1), moderate change (≥ 3.1 to < 5.1 or ≤ -3.1 to > -5.1) or large change (≥ 5.1, ≤ -5.1). The GRCQ evaluated change in respiratory symptoms on a visual analog scale from -7 (worsening) to +7 (improvement). The following algorithm was used to obtain the mean change:
  If the corresponding GRCQ score was in the "no change" group, then change from baseline QOL-B = Observed QOL-B change from baseline score; if > 1, then change from baseline QOL-B score = Observed QOL-B change from baseline score; if < -1, the change from baseline QOL-B score = (-1) * Observed QOL-B change from baseline score.
  Then the mean change from baseline of QOL-B respiratory symptoms score of the minimal change category group is the anchor-based MCID.
Time Frame: Day 0 to Day 28
Population: Participants who were evaluable for MCID and had both GRCQ and QOL-B change values at Day 28 (Visit 4) in any GRCQ domain were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI
Number analyzed (Participants) | 83
units on a scale | 2.9 (10.2)

ADVERSE EVENTS:
Time Frame: Pre-baseline through 70 days
Arm/Group | AZLI
Serious Adverse Events (participants affected / at risk) | 4/89
Other Adverse Events (participants affected / at risk) | 36/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=89)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=89)
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8
Pyrexia (General disorders) | 7
Fatigue (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years